CLINICAL TRIAL: NCT00183105
Title: Hospital-based Brief Intervention for Alcohol Problems
Brief Title: ASAP Study - Hospital-Based Brief Intervention for Alcohol Problems
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Pittsburgh (Other); Boston University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAASaitz12617-ASAP; P60AA013759 (NIH); NIH AA12617
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2007-12

CONDITIONS: Alcohol Dependence; Alcohol Consumption
Keywords: Alcohol; Alcohol abuse; Alcohol dependence; Utilization; Alcohol consumption; Unhealthy alcohol use; Hospitalization; Screening; Brief Intervention; Motivational Interviewing; Randomized trial; Effectiveness; Unhealthy alcohol use (Risky alcohol consumption amounts, problem alcohol use, hazardous alcohol use, alcohol abuse and alcohol dependence)
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Patient Acceptance of Health Care | interventions — Crisis Intervention

INTERVENTIONS:
Behavioral: Brief Intervention (adaptation of motivational interviewing)

SUMMARY:
The objective of this project was to test whether screening and brief intervention for unhealthy alcohol use leads to improved alcohol-related outcomes (such as alcohol consumption and linkage to alcohol assistance) and is cost-effective.

DETAILED DESCRIPTION:
In this study the effectiveness and cost-effectiveness of brief intervention for unhealthy alcohol use in a diverse group of hospitalized medical patients was tested.

We conducted a randomized trial of medical inpatients with the whole spectrum of alcohol problems from risky use through dependence. Subjects in one group received standard care; subjects in the second group received a brief motivational intervention tailored to the severity of his or her alcohol problem. Primary outcomes are alcohol consumption and linkage to alcohol treatment. Additional outcomes include health-related quality of life, health care utilization, alcohol problems, and readiness to change. Costs, and clinical outcomes measured in quality-adjusted life years, a standard metric that allows comparison to other chronic illnesses, will be compared in a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fluent in English or Spanish
* Consume risky amounts of alcohol
* Provide 2 contacts to assist with follow-up
* Have no plans to move from the local area within a year of screening
* Score >21 on Mini-Mental State Examination (no serious cognitive impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2001-02; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Linkage to alcohol assistance
Change in drinks per day

SECONDARY OUTCOMES:
Change in the number of times a subject exceeded per occasion limits
Abstinence (dichotomous)
Change in drinks per day
Drinking risky amounts (dichotomous)
Binge drinking (dichotomous)
Hospitalization
Emergency Department visits
Health related quality of life
Readiness to change alcohol use

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saitz, M.D., M.P.H., Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Kraemer KL, Roberts MS, Horton NJ, Palfai T, Samet JH, Freedner N, Tibbetts N, Saitz R. Health utility ratings for a spectrum of alcohol-related health states. Med Care. 2005 Jun;43(6):541-50. doi: 10.1097/01.mlr.0000163644.97251.14. PMID 15908848
- [Derived] Saitz R, Palfai TP, Cheng DM, Horton NJ, Freedner N, Dukes K, Kraemer KL, Roberts MS, Guerriero RT, Samet JH. Brief intervention for medical inpatients with unhealthy alcohol use: a randomized, controlled trial. Ann Intern Med. 2007 Feb 6;146(3):167-76. doi: 10.7326/0003-4819-146-3-200702060-00005. PMID 17283347